CLINICAL TRIAL: NCT01431339
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy Study to Compare the Efficacy and Safety of Dalbavancin to a Comparator Regimen (Vancomycin and Linezolid) for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: Efficacy and Safety of Dalbavancin for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Durata Therapeutics Inc., an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUR001-302
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2013-12

CONDITIONS: Abscess; Wound Infection; Surgical Site Infection; Cellulitis
MeSH Terms: conditions — Abscess; Wound Infection; Surgical Wound Infection; Cellulitis | interventions — dalbavancin; Vancomycin; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin with possible switch to oral linezolid (Active Comparator)
  Interventions: Drug: Vancomycin/Linezolid
- Dalbavancin (Experimental)
  Interventions: Drug: IV Dalbavancin

INTERVENTIONS:
Drug: IV Dalbavancin — IV Dalbavancin 1000 mg on Day 1 and 500 mg on Day 8
  Arms: Dalbavancin
Drug: Vancomycin/Linezolid — IV Vancomycin (1 gram Q 12 hours or 15mg/Kg Q 12 hours) with optional switch to oral linezolid (600 mg every 12 hours). Total duration of therapy is 10-14 days
  Arms: Vancomycin with possible switch to oral linezolid

SUMMARY:
The primary object is to compare the early clinical efficacy (after 48-72 hours of therapy) of dalbavancin to the comparator regimen (vancomycin with the option to switch to oral linezolid) for the treatment of patients with a suspected or proved gram-positive bacterial skin or skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 - 85 years of age.
2. Signed and dated informed consent document.
3. Major abscess, surgical site infection, traumatic wound infection or cellulitis suspected or confirmed to be caused by Gram-positive bacteria.
4. At least two (2) local signs and symptoms of ABSSSI and at least one (1) systemic sign of infection.
5. Requires a minimum of 3 days of IV therapy.
6. Patient willing and able to comply with study procedures.

Exclusion Criteria:

Patients presenting with any of the following:

1. A contra-indication to any required study drug.
2. Pregnant or nursing females.
3. Sustained shock.
4. Participation in another study of an investigational drug or device within 30 days.
5. Receipt of a systemically or topically administered antibiotic within 14 days prior to randomization, except receipt of a single dose of a short-acting antibacterial drug 3 or more days prior to randomization.
6. Infection due to a dalbavancin or vancomycin-resistant organism.
7. Evidence of meningitis, necrotizing fasciitis, gas gangrene, gangrene, septic arthritis, osteomyelitis, and/or endovascular infection.
8. Exclusively gram-negative bacterial or a fungal ABSSSI.
9. Venous catheter infection.
10. Infection of a diabetic foot ulcer or a decubitus ulcer.
11. Device-related infections.
12. Gram-negative bacteremia.
13. Infected burns.
14. Infected limb with critical ischemia.
15. Superficial/simple skin and skin structure infections.
16. Concomitant condition requiring non-study antibacterial therapy.
17. ABSSSI requiring therapy for longer than 14 days.
18. Adjunctive therapy with hyperbaric oxygen.
19. More than 2 surgical interventions for ABSSSI anticipated.
20. Chronic inflammatory condition precluding assessment of clinical response.
21. Absolute neutrophil count < 500 cells/mm3.
22. Human immunodeficiency virus (HIV) infection with a CD4 cell count < 200 cells/mm3.
23. Recent bone marrow transplant, > 20 mg prednisolone per day (or equivalent) or receiving immunosuppressant drugs after organ transplantation.
24. Regular, chronic antipyretic use in patients unable to modify during the first three days of study drug therapy.
25. Life expectancy less than 3 months.
26. Conditions that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results.
27. Prior participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunne, MD, Study Director — Durata Therapeutics Inc., an affiliate of Allergan plc
Locations (122):
- United States (30):
  - Durata Clinical Site, Montgomery, Alabama
  - Durata Clinical Site, Anaheim, California
  - Durata Clinical Site, Buena Park, California
  - Durata Study Site, Chula Vista, California
  - Durata Clinical Site, Long Beach, California
  - Durata Study Site, Los Angeles, California
  - Durata Study Site, Norwalk, California
  - Durata Study Site, Oxnard, California
  - Durata Study SIte, San Diego, California
  - Durata Study Site, Stockton, California
  - Durata Clinical Site, Boyton Beach, Florida
  - Durata Clinical Site, Fort Meyers, Florida
  - Durata Clinical Site, Miami, Florida
  - Durata Study Site, Orlando, Florida
  - Durata Clinical Site, Saint Cloud, Florida
  - Durata Clinical Site, Augusta, Georgia
  - Durata Study Site, Columbus, Georgia
  - Durata Clinical Site, Chicago, Illinois
  - Durata Study Site, Baton Rouge, Louisiana
  - Durata Study Site, New Orleans, Louisiana
  - Durata Study Site, Shreveport, Louisiana
  - Durata Study Site, Zachary, Louisiana
  - Durata Study Site, Las Vegas, Nevada
  - Durata Study Site, Springfield, Ohio
  - Durata Study Site, Philadelphia, Pennsylvania
  - Durata Study Site, Austin, Texas
  - Durata Clinical Site, Austin, Texas
  - Durata Clinical Site, Houston, Texas
  - Durata Study Site, Richmond, Texas
  - Durata Study Site, Middleton, Wisconsin
- Bulgaria (4):
  - Durata Study Site, Pleven
  - Durata Study Site, Plovdiv
  - Durata Study Site, Sevlievo
  - Durata Study Site, Sofia
- Estonia (4):
  - Durata Study Site, Kohtla-Järve
  - Durata Clinical Site, Kohtla-Järve
  - Durata Clinical Site, Tallinn
  - Durata Study Site, Tartu
- Hungary (7):
  - Durata Study Site, Budapest
  - Durata Clinical Site, Budapest
  - Durata Study Site, Debrecen
  - Durata Clinical Site, Kaposvár
  - Durata Clinical SIte, Pécs
  - Durata Clinical Site, Szeged
  - Durata Study Site, Veszprém
- Israel (7):
  - Durata Clinical Site, Haifa
  - Durata Study Site, Jerusalem
  - Durata Clinical Site, Kfar Saba
  - Durata Clinical Site, Petah Tikva
  - Durata Study Site, Petah Tikva
  - Durata Clinical Site, Ramat Gan
  - Durata Study Site, Tel Aviv
- Latvia (6):
  - Durata Clinical Site, Daugavpils
  - Durata Clinical Site, Liepāja
  - Durata Study Site, Rēzekne
  - Durata Study Site, Riga
  - Durata Clinical Site, Riga
  - Durata Clinical Site, Ventspils
- Lithuania (5):
  - Durata Clinical Site, Kaunas
  - Durata Clinical Site, Kauno M. Sav
  - Durata Clinical Site, Klaipėda
  - Durata Clinical Site, Šiauliai
  - Durata Clinical Trial, Vilnius
- Romania (8):
  - Durata Study Site, Bucharest
  - Durata Clinical Site, Bucharest
  - Durata Clinical Trial, Bucharest
  - Durata Clinical Site, Burcharest
  - Durata Study Site, Cluj-Napoca
  - Durata Study Site, Constanța
  - Durata Study Site, Târgu Mureş
  - Durata Clinical Site, Timișoara
- Russia (11):
  - Durata Clinical Site, Vsevolozhsk, Leningradskaya Oblast'
  - Durata Study Site, Vsevolozhsk, Leningradskaya Oblast'
  - Durata Study Site, Moscow
  - Durata Clinical Site, Moscow
  - Durata Study Site, Petrozavodsk
  - Durata Clinical Site, Saint Petersburg
  - Durata Clinical Site, Smolensk
  - Durata Study Site, Tomsk
  - Durata Clinical Site, Tver'
  - Durata Clinical Site, Volgograd
  - Durata Clinical Site, Yaroslavl
- Slovakia (4):
  - Durata Clinical Site, Banská Bystrica
  - Durata Clinical Site, Levice
  - Durata Clinical Site, Nitra
  - Durata Clinical Site, Svidník
- South Africa (11):
  - Durata Study Site, KwaZulu, Durban
  - Durata Study Site, KwaZulu-Natal, Ladysmieth
  - Durata Study Site, Mpumalanga, Middleburg
  - Durata Study Site, Mpekweni, Paarl
  - Durata Study Site, Western Cape, Paarl
  - Durata Clinical Site, Gauteng, Pretoria
  - Durata Study Site, Gauteng, Soweto
  - Durata Study Site, Johannesburg
  - Durata Study Site, Port Elizabeth
  - Durata Clinical Site, Pretoria
  - Durata Study Site, Thabazimbi
- South Korea (8):
  - Durata Clinical Site, Jung Gu, Daegu
  - Durata Clinical Site, Ansan
  - Durata Study Site, Daejeon
  - Durata Study Site, Gwangju
  - Durata Clinical Site, Incheon
  - Durata Clinical Site, Kangwon-do
  - Durata Study Site, Seoul
  - Durata Clinical Site, Seoul
- Taiwan (6):
  - Durata Study Site, Tainan, Fukien
  - Durata Study Site, Kaohsiung City
  - Durata Clinical Site, Taichung
  - Durata Clinical Site, Taipai
  - Durata Study Site, Taipei
  - Durata Study Site, Yung Kang City
- Ukraine (11):
  - Durata Study Site, Cherkasy
  - Durata Study Site, Dnipropetrovsk
  - Durata Study Site, Donetsk
  - Durata Clinical Site, Ivano-Frankivsk
  - Durata Study Site, Ivano-Frankivsk
  - Durata Study Site, Kharkiv
  - Durata Clinical Site, Kyiv
  - Durata Study Site, Kyiv
  - Durata Study Site, Lviv
  - Durata Study Site, Uzhhorod
  - Durata Study Site, Zaporizhia

REFERENCES:
- [Derived] Gonzalez PL, Rappo U, Akinapelli K, McGregor JS, Puttagunta S, Dunne MW. Outcomes in Patients with Staphylococcus aureus Bacteremia Treated with Dalbavancin in Clinical Trials. Infect Dis Ther. 2022 Feb;11(1):423-434. doi: 10.1007/s40121-021-00568-7. Epub 2021 Dec 14. PMID 34905144
- [Derived] Boucher HW, Wilcox M, Talbot GH, Puttagunta S, Das AF, Dunne MW. Once-weekly dalbavancin versus daily conventional therapy for skin infection. N Engl J Med. 2014 Jun 5;370(23):2169-79. doi: 10.1056/NEJMoa1310480. PMID 24897082

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalbavancin | Vancomycin With Possible Switch to Oral Linezolid
Started | 371 | 368
Safety Population | 368 | 367
Completed | 332 | 333
Not Completed | 39 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin | Vancomycin With Possible Switch to Oral Linezolid | Total
Number analyzed (Participants) | 371 | 368 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (16.54) | 51.4 (16.16) | 50.2 (16.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 167 | 315
  Male | 223 | 201 | 424

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Efficacy
Description: Clinical response at 48-72 hours post study drug initiation, based on measurements of acute bacterial skin and skin structure infections (ABSSSI) lesion size and temperature
Time Frame: After 48-72 hours of therapy
Population: The ITT population consisted of all randomly assigned patients regardless of whether or not they received study drug.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin With Possible Switch to Oral Linezolid
Number analyzed (Participants) | 371 | 368
participants
  Clinical Responder | 285 | 288
  Clinical Non-Responder | 86 | 80
Statistical Analysis 1: Comparison: Dalbavancin vs Vancomycin With Possible Switch to Oral Linezolid; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis test is a one-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the 95% CI for the difference in response rates in the ITT population is greater than -10% the NI of dalbavancin to vancomycin/linezolid will be concluded; Difference in Proportions = -1.5, 95% CI [-7.4 to 4.6] — Confidence intervals were adjusted for fever at baseline

2. Secondary Outcome: Clinical Status
Description: Compare the clinical efficacy at end of treatment visit of dalbavancin to the comparator regimen based on lesion size, local signs, temperature and receipt of other therapy
Time Frame: End of Treatment Visit (Day 14-15)
Population: Clinical Evaluable Population based on certain inclusion/exclusion criteria, length of study therapy, concomitant antibacterials, concomitant surgical procedure and non-missing data.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin With Possible Switch to Oral Linezolid
Number analyzed (Participants) | 324 | 302
participants
  Clinical Succcess | 303 | 280
  Clinical Failure | 21 | 22

3. Secondary Outcome: >= 20% Reduction in Lesion Area
Description: Clinical response at 48-72 hours post study drug initiation, based on measurements of acute bacterial skin and skin structure infections (ABSSSI) lesion size
Time Frame: 48-72 hours after the initiation of study therapy
Population: The ITT population consisted of all randomly assigned patients regardless of whether or not they received study drug.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin With Possible Switch to Oral Linezolid
Number analyzed (Participants) | 371 | 368
participants
  Clinical Responder | 325 | 316
  Clinical Non-Responder | 46 | 52

4. Secondary Outcome: Clinical Status
Description: Compare the clinical efficacy at the short term follow-up visit of dalbavancin to the comparator regimen based on lesion size, local signs temperature and receipt of other therapy
Time Frame: Follow-Up Visit (day 28)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin With Possible Switch to Oral Linezolid
Number analyzed (Participants) | 294 | 272
participants
  Clinical Success | 283 | 257
  Clinical Failure | 11 | 15

ADVERSE EVENTS:
Time Frame: Begins from the time that the patient provides informed consent through the last follow up visit, Day 70. Any SAE occurring any time after the reporting period must be promptly reported if a causal relationship to investigational product is suspected.
Description: Adverse events were analyzed in the safety population which is defined as all patients in the ITT population who received at least 1 dose of dalbavancin or vancomycin (active) study drug.
Arm/Group | Dalbavancin | Vancomycin With Possible Switch to Oral Linezolid
Serious Adverse Events (participants affected / at risk) | 12/368 | 14/367
Other Adverse Events (participants affected / at risk) | 29/368 | 28/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalbavancin (N=368) | Vancomycin With Possible Switch to Oral Linezolid (N=367)
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Sudden death (General disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Gangrene (Infections and infestations) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalbavancin (N=368) | Vancomycin With Possible Switch to Oral Linezolid (N=367)
Nausea (Gastrointestinal disorders) | 15 | 15
Headache (Nervous system disorders) | 11 | 9
Vomiting (Gastrointestinal disorders) | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will provide Durata an opportunity to review any proposed publication or other type of disclosure at least 30 days before they are submitted. If any patent action is required to protect intellectual property rights, the Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days. If the study is part of a multi-center study, the Investigator agrees that the first publication is to be a joint publication covering all centers.